CLINICAL TRIAL: NCT03021408
Title: Evaluation of the Effectiveness of Three Different Approaches for the Rehabilitation of Gait in Patients With Parkinson's Disease: Treadmill Versus Treadmill-plus Versus Virtual Reality
Brief Title: Effectiveness of Different Approaches for the Rehabilitation of Gait in Patients With Parkinson's Disease
Acronym: Tr-T-VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OGZonaMP-PD Gait Rehab
Record Dates: First submitted 2017-01-07; First posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: PD; Gait Dysfunction, Neurologic; Rehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MIRT + Treadmill (Experimental): In the context of MIRT, the gait training in this group will be performed by using a treadmill without cues.
  Interventions: Other: MIRT + Treadmill
- MIRT + Treadmill Plus (Experimental): In the context of MIRT, the gait training in this group will be performed by using a treadmill with visual and auditory cues.
  Interventions: Other: MIRT + Treadmill Plus
- MIRT + Virtual Reality (Experimental): In the context of MIRT, the gait training in this group will be performed by using Virtual Reality with enhanced perceptions (visual, auditory, and haptic inputs).
  Interventions: Other: MIRT + Virtual Reality

INTERVENTIONS:
Other: MIRT + Treadmill — PD patients will undergo a 4-week MIRT. All patients in the MIRT+Treadmill Plus group will undergo 10-minutes treadmill training twice per day, 5 times a week, for 4 weeks.
  Arms: MIRT + Treadmill
Other: MIRT + Treadmill Plus — PD patients will undergo a 4-week MIRT. All patients in the MIRT+Treadmill Plus group will undergo 10-minutes treadmill-plus training (with visual and auditory cues) twice per day, 5 times a week, for 4 weeks.
  Arms: MIRT + Treadmill Plus
Other: MIRT + Virtual Reality — PD patients will undergo a 4-week MIRT. All patients in the MIRT+Virtual Reality (VR) group will undergo 10-minutes VR training with enhanced perceptions (visual, auditory, and haptic inputs), twice per day, 5 times a week, for 4 weeks.
  Arms: MIRT + Virtual Reality

SUMMARY:
Evaluation of the effectiveness of three different approaches for the rehabilitation of gait in patients with PD within a multidisciplinary, intensive rehabilitation treatment (MIRT).

DETAILED DESCRIPTION:
Gait disorders represent one of principal hallmark of Parkinson's disease (PD). Typically, PD patients demonstrate reduced stride length and walking speed during free ambulation, while double support duration and cadence rate are increased. Gait disorders are generally poorly responsive to dopaminergic treatments and are related to reduced quality of life and augmented risk of falls. Different rehabilitation techniques based on compensatory and learning strategies, which principally exploit the use of cues to bypass the defective basal ganglia and to ameliorate performance through practice, have been demonstrated to be effective in improving gait in patients with PD. Cueing techniques represent the central core for the rehabilitation of parkinsonian gait. In this context, it has been demonstrated that treadmill training can improve gait performance in PD patients. It probably acts as an external cue exerting a normalizing effect on the spatiotemporal gait parameters and leading to an enhanced gait rhythmicity and a reduced gait variability. The use of a treadmill with visual and auditory cues (treadmill-plus) seems to lead to a better improvement in gait parameters when compared to treadmill alone. Recently, the application of virtual reality (VR) has been introduced in the rehabilitation of PD. The use of VR is based on the interaction of the person with a virtual environment with the aim to promote motor learning through enhanced perceptions (visual, auditory, and haptic inputs).

It has been widely demonstrated that a multidisciplinary, intensive, goal-based, motor-cognitive and aerobic treatment (MIRT), specifically designed for PD patients, provide parkinsonians with motor and functional benefits. Nevertheless, the contribution provided by treadmill, treadmill-plus and VR on gait parameters has not been previously addressed within MIRT.

This study aims at investigating the superiority or the non-inferiority of these different devices in improving gait in PD patients in the context of MIRT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "probable" idiopathic Parkinson's disease according to Gelb et al (Gelb, 1999);
* Mild to moderate stage of disease (stage 2-3) according to Hoehn & Yahr scale;
* Ability to walk on treadmill;
* Visual and hearing capacity sufficient to perceive the cues;
* No cognitive impairment (Mini-Mental State Examination score ≥ 26);
* Stable pharmacological treatment since 2 weeks before admission and during rehabilitation;

Exclusion Criteria:

* Diagnosis of atypical or vascular Parkinsonism;
* Occurrence of cardiovascular, orthopaedic, peripheral nerves, musculoskeletal and vestibular disorders which could affect patient's locomotion or balance;
* Neuropsychiatric disturbances;
* Severe dyskinesia;
* Severe freezing of gait;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
6-minute walking test (6MWT) | 4 weeks
  Patient is first familiarized with the test by letting him/her go once forward and backward along a straight 15-m line on the ground in a gymnasium. Then, after 15 minutes rest, he/she is instructed to walk from end to end of the line for 6 minutes and to cover as much distance as possible. No encouragement is offered during the test and no cues are used.

SECONDARY OUTCOMES:
Average length of right and left steps | 4 weeks
  The average length of right and left steps (expressed in centimetres and calculated by averaging the length of all the right steps and left steps, respectively).
Coefficient of variance | 4 weeks
  coefficient of variance (CoV) of both right and left steps (which expresses the amount of variation occurring between footfalls).
Step cycle | 4 weeks
  Step cycle (cycle/s), calculated by averaging the step cycles during the exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Frazzitta Giuseppe, MD, Study Director — "Moriggia-Pelascini" Hospital
Locations (1):
- "Moriggia-Pelascini" Hospital, Gravedona Ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No